CLINICAL TRIAL: NCT05050877
Title: Risk Factors and Prognosis of Adverse Cardiovascular and Kidney Events After Coronary Intervention - Cardiorenal ImprovemeNt Registry II
Brief Title: Risk Factors and Prognosis of Adverse Cardiovascular and Kidney Events After Coronary Intervention II
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Maoming Hospital Affiliated to Southern Medical University (Unknown); Shenzhen People's Hospital (Other); Yangjiang People's Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Chen, Director, Guangdong Provincial People's Hospital
Other Study IDs: 2019-555H-2
Record Dates: First submitted 2021-09-09; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cardio-Renal Syndrome; Coronary Angiography; Coronary Artery Disease; Kidney Diseases; Metabolic Syndrome
Keywords: contrast-induced acute kidney injury; contrast medium; creatinine clearance; coronary angiography; chronic kidney disease; Adverse Cardiovascular and Kidney Events
MeSH Terms: conditions — Cardio-Renal Syndrome; Coronary Artery Disease; Kidney Diseases; Metabolic Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary angiography: The investigators recruit all consecutive patients who were undergoing coronary angiography or percutaneous coronary intervention.

SUMMARY:
As a multi-center, retrospective observation study in southern China, this study included the main study population of patients who underwent coronary angiography at 5 hospitals from Guangzhou, Shenzhen, Yangjiang, Maoming and Longyan from January 2000 to Decemeber 2020. The hospitalization information was collected in the form of direct derivation of the case, and cardiac and renal adverse events were collected through outpatient system. Data on all-cause death were obtained from the Guangdong Provincial Public Security and matched to the electronic Clinical Management System of the Guangdong Provincial People's Hospital records.

DETAILED DESCRIPTION:
This is a multi-center, retrospective observation study collecting data on 184855 coronary angiography patients from January 2000 to Decemeber 2020. Data regarding demographic information, admission diagnoses and history of present illness, biomarkers and details on preventive hydration and medications will be collected. The primary endpoint of this study is Adverse Cardiovascular and Kidney Events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to CAG or PCI;

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators reviewed all consecutive patients who were undergoing coronary angiography.
Sampling Method: Probability Sample
Enrollment: 184855 (Actual)
Dates: Start 2000-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Contrast-Induced Acute Kidney Injury (CI-AKI 0.3) | 48 hours
  defined as a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure

SECONDARY OUTCOMES:
Cystatin C based CI-AKI (CI-AKI cyc) | 24-48 hours
  Cystatin C based CI-AKI, defined as a ≥10% absolute increase in serum cystatin C during the first 24 hours after the procedure and and a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure.mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure.
The change of eGFR, calculate based on CrCl and serum cystatin C | 48-72 hours
  The eGFR creatinine-cystatin C was calculated by the 2012 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) cystatin C equation: 135 *min(Scr/κ, 1)α * max(Scr/κ, 1)-0.601 * min(Scys/0.8, 1)-0.375 * max (Scys/0.8, 1)-0.711 * 0.995Age [* 0.969 if female] [* 1.08 if black], where Scr is serum creatinine, Scys is serum cystatin C, κ is 0.7 for females and 0.9 for males, α is -0.248 for females and -0.207 for males, min indicates the minimum of Scr/κ or
  1, and max indicates the maximum of Scr/κ or 1.

OTHER OUTCOMES:
Contrast-induced Persistent kidney injury (CI-PKI) | 3 months
  Serum creatinine was measured by endpoint colorimetry or enzymatic assays. CI-PKI was defined as residual impairment of renal function indicated by a ≥ 25% reduction in creatinine clearance at 3 months in comparison with baseline. comparison with baseline.
Incidence of major adverse cardiovascular events | 3-12months
  all-cause mortality (cardiovascular and noncardiovascular) and cardiovascular events.
Follow-up major adverse cardiovascular and clinical events | 3-12months
  We will follow up the patients by telephone and outpatient service to know the one year all-cause mortality (cardiovascular and noncardiovascular) and cardiovascular events.
All-cause mortality | From the hospital admission, and up to 10 years
  Died for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD,PhD, Study Director — Guangdong Cardiovascular Institute,Guangdong Provincial People's Hospital; Shiqun Chen, MS, Study Director — Guangdong Cardiovascular Institute,Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng L, Chen H, Xu Q, Han K, Liu J, Chen S, Deng J, Tian L, Li Z, Lu X, Liu Y, Liang Y. The High-Sensitivity C-Reactive Protein to High-Density Lipoprotein Cholesterol Ratio and the Risk of Contrast-Induced Acute Kidney Injury in Patients Undergoing Percutaneous Coronary Intervention. Rev Cardiovasc Med. 2024 Sep 23;25(9):338. doi: 10.31083/j.rcm2509338. eCollection 2024 Sep. PMID 39355575
- [Derived] Zhou Z, Qiao L, Ling Y, He Y, Chang T, Lu H, Yu S, Liu J, Guo W, Chen S, Liu Y, Chen J. Intermediate Hyperglycemia Increases the Risk of All-Cause Mortality in Premature Coronary Artery Disease Patients Undergoing Percutaneous Coronary Intervention. Rev Cardiovasc Med. 2023 Dec 13;24(12):352. doi: 10.31083/j.rcm2412352. eCollection 2023 Dec. PMID 39077077
- [Derived] Xie Y, Xu X, Wang D, Zhou Y, Kang Y, Lai W, Lu H, Liu J, Chen S, Xu J, Yan X, Huang X, Liu Y. Fibrinogen-to-Albumin Ratio and Long-Term Mortality in Coronary Artery Disease Patients with Different Glucose Metabolism Status. Rev Cardiovasc Med. 2023 Nov 16;24(11):317. doi: 10.31083/j.rcm2411317. eCollection 2023 Nov. PMID 39076427
- [Derived] Wu W, Jia C, Xu X, He Y, Xie Y, Zhou Y, Lu H, Liu J, Chen J, Liu Y. Impact of Platelet-to-HDL-Cholesterol Ratio on Long-Term Mortality in Coronary Artery Disease Patients with or Without Type 2 Diabetes: Insights from a Chinese Multicenter Cohort. J Inflamm Res. 2024 May 6;17:2731-2744. doi: 10.2147/JIR.S458950. eCollection 2024. PMID 38737110
- [Derived] Jia C, Wu W, Lu H, Liu J, Chen S, Liang G, Zhou Y, Yu S, Qiao L, Chen J, Tan N, Liu Y, Chen J. Fibrinogen to HDL-Cholesterol ratio as a predictor of mortality risk in patients with acute myocardial infarction. Lipids Health Dis. 2024 Mar 25;23(1):86. doi: 10.1186/s12944-024-02071-7. PMID 38528580
- [Derived] Lu J, He Y, Yang Y, Zhong X, Chen S, Wu B, Pan Y, Wang Y, Xiu J, Kang Y, Liu J, Liu Y, Chen S, Chen K, Chen L. Age-Related Effect of Uric Acid on Contrast-Induced Acute Kidney Injury of Patients Undergoing Coronary Angiography. Clin Interv Aging. 2023 Dec 7;18:2053-2061. doi: 10.2147/CIA.S419370. eCollection 2023. PMID 38088947
- [Derived] Liu J, Chen S, Zhou Y, Huang H, Li Q, Liang Y, Dong S, Huang X, Chen L, Zheng X, Meng R, Jia C, Chen J, Tan N, Liu Y. Proportion and number of incident cancer deaths in coronary artery disease. Cancer Med. 2023 Oct;12(19):20140-20149. doi: 10.1002/cam4.6595. Epub 2023 Sep 27. PMID 37754571
- [Derived] Liu J, Chen S, Zhou Y, Zheng X, Meng R, Tan N, Liu Y. Effect of cumulative radiation exposure from Coronary catheterization on lung cancer mortality. BMC Cancer. 2023 Aug 15;23(1):757. doi: 10.1186/s12885-023-11231-4. PMID 37582730
- [Derived] Gao F, Huang Z, Liang J, Kang Y, Ling Y, He Y, Chen J, Hong D, Zhang Z, Xu S, Wang A, Yan X, Liu J, Liu Y, Chen S, Chen J. Association of malnutrition with all-cause and cardiovascular mortality in patients with mild to severe chronic kidney disease undergoing coronary angiography: a large multicenter longitudinal study. Int Urol Nephrol. 2023 Dec;55(12):3225-3236. doi: 10.1007/s11255-023-03566-5. Epub 2023 Apr 27. PMID 37103656